CLINICAL TRIAL: NCT04829266
Title: Effect of Mental Simulations on the Early Mobilization of Patients After Cesarean Section
Brief Title: Mental Simulations and Early Mobilization of Patients After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Anna Prokopowicz, MSc, Principal Investigator, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 05P/12-2017
Record Dates: First submitted 2021-03-23; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Anxiety; Cesarean Section
Keywords: mental simulation; anxiety; verticalization; obstetrics; cesarean section; post-operative care
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- process simulation group (Experimental): an experimental group with process simulation with elements of relaxation
  Interventions: Behavioral: mental simulation
- outcome simulation group (Experimental): an experimental group with outcome simulation with elements of relaxation
  Interventions: Behavioral: mental simulation
- control group (Other): a control group with no process and outcome simulations, but with elements of relaxation
  Interventions: Behavioral: mental simulation

INTERVENTIONS:
Behavioral: mental simulation — Audio recordings with a mental simulation. The women listened to the text using headphones about 10-15 min before verticalization (5 h after arrival in the postoperative room, about 6 h after anesthesia). In each group, the mental training lasted for about 10 min.
  Other Names: The recording of the process simulation included the order to imagine subsequent elements of the process of mobilization.; The recording of the outcome simulation included an optimistic vision of returning to health and fitness.; A fragment of the book "Little Prince" by Antoine de Saint-Exupéry, including an order to imagine the elements of the world as seen through the eyes of the main character

SUMMARY:
Mental simulations can motivate patients for their first verticalization after cesarean section, although perceived anxiety before verticalization may reduce a positive effect of mental simulations.

ELIGIBILITY:
Inclusion Criteria:

* must be qualified to and undergoing delivery using Cesarean section,
* must be undergoing conduction of anesthesia during Cesarean section,
* must be undergoing the analgesic therapy in the postoperative period,
* must be qualified to mobilization by the medical staff,
* must be fluent in Polish in speaking and writing.

Exclusion Criteria:

* any orthopedic dysfunction,
* any neurological dysfunction,
* any psychiatric disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-05-27 (Actual); Study Completion 2018-05-27 (Actual)

PRIMARY OUTCOMES:
willingness to verticalize | Immediately after a single mental simulation
  Percentage of women who were willing to verticalize after listening to the recording. Assessed on a on a six-point scale.
verticalization | Immediately after a single mental simulation
  Percentage of the success of verticalization after listening to the recording.
duration of the first mobilization | Immediately after a single mental simulation
  Time form the start of the measurement was set at getting out of bed from a sitting position, and the end of the measurement was set at the patient's return to bed.

SECONDARY OUTCOMES:
pain level | 3 time points (before and immediately after a single mental simulation, and immediately after verticalization.
  The average pain she experienced during upright standing. Measured with a 10-point numerical rating scale.
anxiety | upon arrival at the recovery room, before and immediately after a single mental simulation.
  Measured with a 10-point numerical rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Prokopowicz, Principal Investigator — Department of Applied Obstetrics, Faculty of Health Sciences, Wroclaw Medical University
Locations (1):
- 2nd Chair and Clinic of Gynecology and Obstetrics, Jan Mikulicz-Radecki University Teaching Hospital in Wrocław, Wrocław, Poland, Wroclaw, Poland

REFERENCES:
- [Derived] Prokopowicz A, Byrka K. Effectiveness of mental simulations on the early mobilization of patients after cesarean section: a randomized controlled trial. Sci Rep. 2021 Nov 22;11(1):22634. doi: 10.1038/s41598-021-02036-1. PMID 34811410